CLINICAL TRIAL: NCT00486785
Title: Sexuality And Management of Benign Prostatic Hyperplasia With Alfuzosin 10mg Once Daily (XATRAL OD 10mg), Open, 24-week Study
Brief Title: SAMBA: Sexuality And Management of Benign Prostatic Hyperplasia With Alfuzosin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALFUS_L_01667
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — Alfuzosin 10mg Once Daily for 24 weeks

SUMMARY:
Primary Objective:

* To assess the sexual function improvement from baseline to the end of treatment (Week 24 or premature withdrawal (PW)) with XATRAL 10mg OD.

Secondary Objective:

* To evaluate the association between Lower Urinary Tract Symptoms (LUTS) severity and sexual disorders,
* To compare the improvement in sexual function, urinary symptoms and Quality of Life among the different regions,
* To correlate MSHQ (Male Sexual Health Questionnaire) and IIEF-5 (the 5-Item version of the International Index of Erectile Function),
* To assess the onset of action of XATRAL 10mg OD,
* To assess the peak flow rate improvement (Qmax),
* To assess the safety and the tolerability of XATRAL 10mg OD.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from moderate to severe lower urinary tract symptoms (LUTS), suggestive of symptomatic Benign Prostatic Hyperplasia (BPH),
* Patients with an I-PSS total score ≥ 8,
* Patients sexually active

Exclusion Criteria:

* Known history of hepatic or severe renal insufficiency, unstable angina pectoris, concomitant threatening-life condition.
* Previous prostate surgery, minimally invasive procedure within 6 months prior to inclusion. Planned prostate biopsy, prostate surgery or minimally invasive procedure during the whole study period.
* Active urinary tract infection or prostatitis, neuropathic bladder, a diagnosed prostate cancer.
* Patients having received 5α-reductase inhibitors or LUTS related phytotherapy within 6 months prior to inclusion, or α1-blockers within 30 days prior to inclusion. Patients receiving any treatment for erectile dysfunction (i.e. phosphodiesterase-5 inhibitors) at inclusion.
* History of postural hypotension or syncope.
* Known hypersensitivity to alfuzosin.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to the end of treatment in the Male Sexual Health Questionnaire(MSHQ) for sexual function. | 24 weeks
Evaluation of adverse events, vital signs (blood pressure and heart rate), PSA (Prostate-specific antigen; mandatory at baseline and optional at the end of treatment) and serum creatinine assessment (optional at baseline and at the end of treatment) | 24 weeks

SECONDARY OUTCOMES:
- Mean change from baseline to 4, 12, and 24 weeks of treatment in MSHQ in the ejaculation score - Mean change from baseline to 4, 12 and 24 weeks of treatment in MSHQ ejaculation questions, in the erection questions and sexual activity and desire | 24 weeks
- Mean change from baseline to week 1 in I-PSS total score and sub-scores (objective onset of action) - Onset of action based on patient perception (questionnaire at Week 1) | 24 weeks
-Mean change from baseline to 4,12 and 24 weeks of treatment in the I-PSS total score and in the Quality of Life -QOL Mean change from baseline to 4, 12 and 24 weeks of treatment in the I-PSS total score and in the Quality of Life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Ruiz, MD, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, Quito, Ecuador
- Sanofi-Aventis, Guatemala City, Guatemala
- Sanofi-Aventis, México, Mexico